CLINICAL TRIAL: NCT04744285
Title: Effects of Filter Ventilation and Ventilation Information on Product Use Behaviors in Cigarette Smokers (COMET 2 3 1)
Brief Title: Effects of Filter Ventilation and Ventilation Information on Product Use Behaviors in Cigarette Smokers
Acronym: COMET 2 3 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 757820; P01CA217806 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cigarette Smoking-Related Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1 (normal cigarettes) (Active Comparator): Participants receive regular package cigarettes for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.
  Interventions: Other: Cigarette packaging; Other: Data capture; Other: Questionnaire administration
- Condition II (cigarettes with neutral message) (Experimental): Participants receive cigarettes with neutral message "Nothing about this product's color or name means that it will protect a smoker from the health risks of smoking" on package for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.
  Interventions: Other: Cigarette packaging; Other: Data capture; Other: Questionnaire administration
- Condition III (cigarettes with compensation message) (Experimental): Participants receive cigarettes with compensation message "This product has a ventilated filter. Filter vents increase how deeply a smoker inhales without them knowing, which can increase the health risks of smoking" on package for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection
  Interventions: Other: Cigarette packaging; Other: Data capture; Other: Questionnaire administration
- Condition IV cigarettes with blocking message (Experimental): Participants receive cigarettes with blocking message "This product has a ventilated filter. Be sure not to block the vent holes with your fingers or lips, which can increase the health risks of smoking" for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection
  Interventions: Other: Cigarette packaging; Other: Data capture; Other: Questionnaire administration

INTERVENTIONS:
Other: Cigarette packaging — receive normal packet cigarette
Other: Data capture — Attend video sessions
Other: Questionnaire administration — Ancillary studies

SUMMARY:
This clinical trial collects data to see how filter ventilation and ventilation information affects product use behaviors in cigarette smokers. Providing ventilation information on the cigarette package may affect smokers' rating of product appeal, perceptions of health risk, and changes in cigarette consumption.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess how adding messaging to cigarette packages about filter vents and filters influences respondents awareness of filter ventilation, beliefs about the function of filter vents and filters, smoking behavior, ratings of cigarette satisfaction, smoking topography, exposure to nicotine and carbon monoxide, perceptions about the risk of smoking, and intention to stop smoking.

OUTLINE: Participants are randomized to 1 of 4 conditions.

CONDITION I: Participants receive regular package cigarettes for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.

CONDITION II: Participants receive cigarettes with neutral message "Nothing about this product's color or name means that it will protect a smoker from the health risks of smoking" on package for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.

CONDITION III: Participants receive cigarettes with compensation message "This product has a ventilated filter. Filter vents increase how deeply a smoker inhales without them knowing, which can increase the health risks of smoking" on package for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.

CONDITION IV: Participants receive cigarettes with blocking message "This product has a ventilated filter. Be sure not to block the vent holes with your fingers or lips, which can increase the health risks of smoking" for 2 weeks. Participants attend 3 video sessions over 0.5 hour each at baseline, 1, and 2 weeks respectively for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-69 years old
* Currently smoking daily, at least 5 cigarettes per day, for the past year:

  * Primarily using factory-made filtered cigarettes
* Fair and above self-rated physical health (self-rated)
* Fair and above self-rated mental health (self-rated)
* Not planning to quit smoking in the next 30 days
* Able to converse, read, and write in English
* Access to smartphone (e.g., iPhone, Android) for Ecological Momentary Assessment (EMA) component
* Access to a smartphone/tablet/computer with video capabilities and internet access for remote videoconferencing (EMA check-ins)

  * Alcohol Use Disorders Identification Test (AUDIT)-C <7 (i.e., no problematic alcohol consumption)
  * Cannibis use less than or equal to 5 days in the past month
  * No other illegal drug use in the past month (allow for prescription)
* Not pregnant or breastfeeding or planning to become pregnant during the study period
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Age < 21 or > 69
* Using roll-your-own cigarettes or usual brand of cigarettes is unfiltered
* Planning to quit smoking in the next 30 days
* Adults unable to consent
* Minors (any persons under age 21)
* Prisoners
* Poor physical health by self-report
* Poor mental health by self-report:

  * Exclude Dx psychosis, Dx bipolar, K6 score indicating serious psychological distress
  * AUDIT-C score >=7 (i.e. problematic alcohol consumption)
  * Cannabis use >5 days in past month
* Other illegal drug use in past month
* Pregnant or breastfeeding by self-report
* No access to smartphone or videoconferencing

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
Started | 31 | 29 | 33 | 22
Completed | 30 | 28 | 31 | 21
Not Completed | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: There were 5 patients that withdrew prior to any study assessments and no data were recorded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message | Total
Number analyzed (Participants) | 30 | 28 | 31 | 21 | 110
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 0 | 0 | 0 | 0 | 0
  >= 18 years old | 30 | 28 | 31 | 21 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 19 | 19 | 83
  Male | 7 | 6 | 12 | 2 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 28 | 31 | 21 | 110

OUTCOME MEASURES:

1. Primary Outcome: Subjective Questionnaires of Product Evaluation
Description: Will be assessed by Duke Sensory Scale. A 9 item questionnaire with nine items that assess participants' sensory experience All questions are rated on a 7-point Likert scale (with 1 meaning -not at all to 7 - meaning extremely).
Time Frame: At 2 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
Number analyzed (Participants) | 30 | 28 | 31 | 21
units on a scale
  How much did you like the puffs you just took? | 4.27 [1 to 7] | 3.86 [1 to 7] | 4.16 [1 to 7] | 4.9 [1 to 7]
  How satisfying were the puffs you just took? | 4.27 [1 to 7] | 3.82 [1 to 7] | 4.35 [1 to 7] | 4.95 [1 to 7]
  How high in nicotine do you think the puffs were? | 4.33 [1 to 7] | 4.11 [1 to 7] | 4.65 [1 to 7] | 4.43 [1 to 7]
  How similar to your own brand were the puffs? | 3.33 [1 to 7] | 3.54 [1 to 7] | 3.77 [1 to 7] | 3.33 [1 to 7]
  Strength of puffs on tongue | 4.03 [1 to 7] | 3.86 [1 to 7] | 3.61 [1 to 7] | 3.76 [1 to 7]
  Strength of puffs in nose | 3.4 [1 to 7] | 3.21 [1 to 7] | 3.03 [1 to 7] | 2.95 [1 to 7]
  Strength of puffs in back of mouth and throat | 4.1 [1 to 7] | 3.54 [1 to 7] | 4.13 [1 to 7] | 4.14 [1 to 7]
  Strength of puffs in windpipe | 4.13 [1 to 7] | 3.61 [1 to 7] | 4.0 [1 to 7] | 4.19 [1 to 7]
  Strength of puffs in chest | 4.07 [1 to 7] | 3.32 [1 to 7] | 3.84 [1 to 7] | 4.10 [1 to 7]

2. Primary Outcome: Readiness to Quit
Description: Will be assessed by contemplation ladder. This is a 0 to 10 scale, where 0 indicates no willingness/readiness to quit and 10 indicates willing/ready to quit immediately.
Time Frame: At 2 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
Number analyzed (Participants) | 30 | 28 | 31 | 21
score on a scale | 6.27 [1 to 10] | 5.79 [1 to 10] | 6.58 [1 to 10] | 6.24 [1 to 10]

3. Primary Outcome: Withdrawal
Description: Will be assessed by Minnesota Tobacco Withdrawal Scale - a 15 item question scale - with scale of 0 -4, 0=Not at all - 4=Severe. A total score is obtained by summing all 15 items.
Time Frame: At 2 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
Number analyzed (Participants) | 30 | 28 | 31 | 21
score on a scale | 13.2 [1 to 45] | 12.3 [1 to 45] | 8.8 [1 to 45] | 13.9 [1 to 45]

4. Secondary Outcome: Level of Exhaled Carbon Monoxide (CO)
Description: level of CO measured in exhaled breath after a 15 seconds breathhold
Time Frame: At 2 weeks
Population: This outcome data was only measured on a random subset of participants.
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
Number analyzed (Participants) | 6 | 8 | 8 | 8
parts per million | 21.3 (11.0) | 15.0 (10.7) | 22.6 (16.6) | 27.6 (33.6)

ADVERSE EVENTS:
Time Frame: 2 weeks after study enrollment.
Arm/Group | Condition 1 (Normal Cigarettes) | Condition II (Cigarettes With Neutral Message) | Condition III (Cigarettes With Compensation Message) | Condition IV Cigarettes With Blocking Message
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/31 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/31 | 0/21
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/31 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT04744285/Prot_SAP_002.pdf
  • Informed Consent Form (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04744285/ICF_001.pdf